CLINICAL TRIAL: NCT04791007
Title: A Monocentric Phase I Safety, Acceptability, and Pharmacokinetic Trial of OB-002H Gel Administered Vaginally and Rectally in Open-Label and Randomised, Double- Blind, Placebo-Controlled Cohorts of HIV-1 Seronegative Adults
Brief Title: OB-002H Gel Administered Vaginally and Rectally in HIV-1 Seronegative Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Orion Biotechnology Polska Sp. z o.o. (Industry)
Collaborators: Scope International AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: OB-002H-101
Record Dates: First submitted 2021-02-02; First posted 2021-03-10 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: HIV Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single dose administration (Part 1) (Experimental): the dose of the drug (4g OB-002H (8.0 mg/g)) administrated once vaginally or rectally
  Interventions: Drug: OB-002
- Multidose administration (Part 2) (Experimental): the dose of the drug (4g OB-002H (8.0 mg/g)) or placebo administered vaginally through five consecutive days
  Interventions: Drug: OB-002; Drug: Placebo

INTERVENTIONS:
Drug: OB-002 — vaginal or rectal administration
Drug: Placebo — vaginal or rectal administration
  Arms: Multidose administration (Part 2)

SUMMARY:
This is a monocentric phase I study in open-label and randomized, double-blind, placebo-controlled cohorts of HIV-1 seronegative adults to evaluate the safety, acceptability, and pharmacokinetic of OB-002H Gel administrated vaginally and rectally.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 45 years (inclusive).
2. HIV-1 antibody negative as documented at screening.
3. Understands and agrees to local sexually transmitted infection (STI) reporting requirements.
4. Able and willing to provide written informed consent to take part in the trial.
5. Willing and able to return for a follow-up visit one week after last IMP administration, barring unforeseen circumstances.
6. Of good general health in the opinion of the investigator.
7. Willing to be sexually abstinent (anal and vaginal sex) for 72 hours before and after each visit except Visit 1.
8. No participation in other clinical trials within the last three months prior Visit 1 and throughout the trial.
9. Willing to abstain from inserting any non-trial products for rectal or vaginal application for 72 hours prior to each trial visit.
10. For female participants only:

    1. Using (or willing to use) highly effective (i.e. failure rate <1% per year) methods of contraception for the duration of trial participation. Such methods include combined oral or transdermal hormonal contraception associated with inhibition of ovulation, oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device [IUD] or intrauterine hormone-releasing system [IUS] inserted at least 28 days prior to the Screening Visit, bilateral tubal occlusion, surgical sterilization, successful vasectomisation of male partner or sexually abstinent for the past 90 days and during the trial. If the female participant has female partners only, the method of contraception will be noted as abstinence to heterosexual activities in the trial documentation.
    2. Not pregnant at the screening.
    3. Not breastfeeding at screening nor intending to breastfeed during trial participation per participant report.

    In addition, participants enrolled in the corresponding cohorts must meet the following criteria:
11. Cohorts A1 and B1 only: Willing to stay at the site overnight for two nights.
12. Cohort A2 only: Willing to stay at the site overnight for six nights.
13. Cohort A3 only: Willing to stay at the site overnight from Day 1 to Day 2 and from Day 5 to Day 6 for PK blood sampling.

Exclusion Criteria:

1. Following laboratory findings at screening:

   1. Haemoglobin < 10.0 g/dL
   2. Platelet count < 100 000/mm3
   3. White blood cell count < 2 000 cells/mm3 or > 15 000 cells/mm3
   4. Glomerular filtration rate (GFR) < 60 mL/min/1.73 m2
   5. Alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 2.5× laboratory upper limit of normal (ULN)
   6. Abnormal glucose or protein on urinalysis (UA)
2. Known allergy or intolerance to any of the IMP excipients (sodium sorbate, sodium chloride, acetic acid, natrasol).
3. By participant report at screening: Use of post-exposure prophylaxis (PEP) for HIV exposure, systemic immunomodulatory medications vaginally or rectally administered medications, and vaginally or rectally administered products (including condoms) containing nonoxynol-9 (N-9) within the last four weeks prior to Visit 1.
4. Any significant underlying medical condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make trial participation unsafe, make the individual unsuitable for the trial or unable to comply with the trial requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cardiovascular, immunological or cerebral disease.
5. Abnormalities of the cervical (females only), vaginal (females only), or colorectal mucosa, or significant symptom(s), which in the opinion of the clinician represents a contraindication to protocol-required biopsies (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external haemorrhoids).
6. Suspected or confirmed drug or alcohol abuse.
7. Positive hepatitis B virus (HBV) or hepatitis C virus (HCV) test results. HSV-1 or HSV-2 seropositive diagnosis will only be allowed if no active lesions are present and since treatment is not required.
8. Body mass index (BMI) < 18 or > 30 kg/m2.
9. Previous enrolment to any preceding cohort of this trial.
10. Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.
11. In addition to the criteria listed above, female participants will be excluded if they meet any of the following criteria:

    1. Last pregnancy outcome or gynaecological surgery within 90 days prior to screening
    2. Chronic and/or recurrent symptomatic vaginal candidiasis at screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of OB-002H gel after single- and multiple-dose application based on the number of observed AEs | approximately 5 weeks for single dose and approximately five to seven weeks for multi-dose
  For the primary safety analysis, the number of ≥ Grade 2 AEs, as well as the number and the percentage of participants with corresponding AEs, will be tabulated overall and per cohort, by system organ class (SOC) and by preferred term (PT).
  Additional AE analyses will also tabulate the number of AEs ≥ Grade 2 observed overall, by relationship and by severity. AEs ≥ Grade 2 that lead to discontinuation of trial participation will be tabulated separately. The safety set will be used for the primary safety analysis.

SECONDARY OUTCOMES:
Acceptability | assessment done on the visit conducted 24 hours after IMP administration
  Participants will receive a placebo sample to check and evaluate the OB-002H gel and will be asked to answer the questions in the questionnaire with Likert scale
OB-002 serum concentration at different time points for the calculation of PK parameters (area under the concentration-time curve (AUC). | Serum samples collected within 24 hours after dosing
  In each Part of the trial, the parameters will be summarised descriptively by cohort and treatment arm (Part 2 only: OB-002H and placebo).
OB-002 serum concentration at different time points for the calculation of PK parameters (maximum concentration (Cmax). | Serum samples collected within 24 hours after dosing
  In each Part of the trial, the parameters will be summarised descriptively by cohort and treatment arm (Part 2 only: OB-002H and placebo).
OB-002 serum concentration at different time points for the calculation of PK parameters (time to maximum concentration (tmax). | Serum samples collected within 24 hours after dosing
  In each Part of the trial, the parameters will be summarised descriptively by cohort and treatment arm (Part 2 only: OB-002H and placebo).
OB-002 serum concentration at different time points for the calculation of PK parameters (minimum concentration (Cmin). | Serum samples collected within 24 hours after dosing
  In each Part of the trial, the parameters will be summarised descriptively by cohort and treatment arm (Part 2 only: OB-002H and placebo).
OB-002 serum concentration at different time points for the calculation of PK parameters (concentration half-life (t½). | Serum samples collected within 24 hours after dosing
  In each Part of the trial, the parameters will be summarised descriptively by cohort and treatment arm (Part 2 only: OB-002H and placebo).

OTHER OUTCOMES:
Exploratory | Serum samples collected within 24 hours after dosing (for cohorts with vaginal gel application)
  To assess the drug concentration in the vaginal fluid after OB-002H gel application
Exploratory | Fluid samples collected within 24 hours after dosing (for cohort with rectal gel application)
  To assess the drug concentration in the rectal fluid after OB-002H gel application
Exploratory | Samples collected on baseline and follow up vist (approximately one week after dosing)
  To determine if any changes in vaginal microflora are observed after OB-002H gel application
Exploratory | Samples collected on baseline and follow up vist (approximately one week after dosing)
  To determine if any changes in rectal microflora are observed after OB-002H gel application
Exploratory | Samples collected on baseline and follow up vist (approximately one week after dosing)
  To determine if any changes in cervical histopathology are observed after OB-002H gel application
Exploratory | Samples collected on baseline and follow up vist (approximately one week after dosing)
  To determine changes in rectal histopathology are observed after OB-002H gel application

CONTACTS AND LOCATIONS:
Locations (1):
- BioVirtus Centrum Medyczne Sp. z o.o., Józefów, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGowan IM, Tzakis N, Kosak B, Korczak B, Engstrom J, Tomaszewska-Kiecana M, Hartley O. Evaluation of the Safety, Acceptability, and Pharmacokinetic Profile of a Gel Formulation of OB-002 in Healthy Volunteers. AIDS Res Hum Retroviruses. 2021 Jun;37(6):453-460. doi: 10.1089/AID.2021.0010. Epub 2021 Apr 30. PMID 33749321